CLINICAL TRIAL: NCT07132047
Title: Mulligan Mobilization Sustained Natural Apophyseal Glide Versus Active Release Technique in Cervicogenic Headache
Brief Title: Mulligan SNAG Versus Active Release Technique in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0028
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Cervicogenic Headache
Keywords: Mulligan mobilization; Active release Technique; Cervicogenic headache; physiotherapy; Neck pain; Manual therapy; Sustained natural apophyseal glide SNAG; range of motion, Articular
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Mulligan Mobilization SNAG with Home Exercise (Experimental): Participants in this arm will receive Headache SNAG Mulligan mobilization, a postero-anterior mobilization of the second cervical vertebra sustained for 10-30 seconds to reduce headache intensity. A maximum of six repetitions will be performed if headache reduction occurs during the first application. In addition, participants will follow a home exercise program consisting of C1-C2 self-SNAG in rotation using a towel to apply pressure to the posterior arch of C1 while actively rotating the cervical spine. Each position will be held for 10 seconds and repeated 10 times twice daily. Written instructions will be provided to ensure compliance.
  Interventions: Other: Mulligan Mobilization SNAG with Home Exercise
- Active Release Technique with Home Exercise (Experimental): Participants will receive Active Release Technique (ART) targeting neck and shoulder soft tissues. The program includes sitting chair stretch, Brugger's stretch, wall angles, and doorway stretches for pectoralis major, upper trapezius, and levator scapulae. Additional movements include head and neck retractions and strengthening of rhomboids, deep neck flexors, and serratus anterior through the Kibler squeeze. A home program of neck stretches hold 20 to 30 sec, 3 times and chin tucks hold 5 sec, 10 times for 2 to 3 sets. posture-improving exercises will be performed to relieve tension, improve alignment, and lessen headache symptoms.
  Interventions: Other: Active Release Technique with Home Exercise

INTERVENTIONS:
Other: Mulligan Mobilization SNAG with Home Exercise — This intervention combines manual mobilization and self-exercise. The therapist applies sustained postero-anterior glides to the second cervical vertebra for 10-30 seconds, up to six repetitions if pain decreases. The home program involves C1-C2 self-SNAG with a towel, maintaining end-range rotation for 10 seconds before returning to neutral. Exercises are completed twice daily for 10 repetitions each session. Participants receive illustrated instructions to promote correct execution and compliance.
  Other Names: Mulligan Mobilization SNAG; Self-SNAG Exercise Program
  Arms: 1. Mulligan Mobilization SNAG with Home Exercise
Other: Active Release Technique with Home Exercise — This approach integrates manual soft tissue release with targeted exercise. ART is applied to the neck and shoulder region, focusing on pectoralis major, upper trapezius, and levator scapulae. Exercises include wall angles, doorway stretches, Brugger's stretch, and head/neck retractions. Strengthening activities target rhomboids, deep neck flexors, and serratus anterior. The home routine consists of neck stretches, chin tucks, and postural drills, performed regularly to enhance muscle balance, posture, and headache relief.
  Other Names: Active Release Technique with Cervical and Shoulder Exercise Program; Soft Tissue Release and Postural Exercise
  Arms: Active Release Technique with Home Exercise

SUMMARY:
This study is designed to compare two different manual therapy approaches for individuals with cervicogenic headaches, a type of headache that originates from the neck. Participants will be randomly assigned to one of two groups.

The first group will receive Mulligan mobilization using sustained natural apophyseal glides (SNAG) along with a home program of Mobilization self-SNAG exercises.

The second group will receive the Active Release Technique (ART) combined with a home program of stretching and strengthening exercises for the neck and shoulder muscles. Each participant will attend treatment sessions three times per week for four weeks. Pain levels, headache impact, and neck function will be evaluated at the start, after four weeks of treatment, and again at eight weeks to determine which method provides better outcomes.

DETAILED DESCRIPTION:
Cervicogenic headache is a form of secondary headache caused by dysfunction in the cervical spine. It is often associated with neck pain, restricted mobility, and limitations in daily activities. Manual therapy, combined with targeted exercises, is frequently used in rehabilitation to reduce pain and improve neck function. This randomized controlled trial aims to compare the effectiveness of Mulligan mobilization with sustained natural apophyseal glides (SNAG) versus the Active Release Technique (ART) in the treatment of cervicogenic headache.

Group A - Mulligan Mobilization SNAG and Home Exercise:

Participants in this group will receive the Headache SNAG technique, which involves a gentle, sustained postero-anterior glide of the second cervical vertebra for 10 to 30 seconds to help reduce headache intensity. If relief is noted, up to six repetitions may be performed. In addition, each participant will be prescribed a home program consisting of C1-C2 self-SNAG rotation using a towel to apply pressure on the posterior arch of C1 during active cervical rotation. The exercise will be completed twice daily, with 10 repetitions per session. Written instructions will be given to ensure correct performance and better compliance.

Group B - Active Release Technique and Home Exercise Program:

Participants allocated to this group will receive the Active Release Technique (ART), a hands-on treatment aimed at releasing tight muscles and improving soft tissue mobility. During ART, controlled pressure is applied to specific muscles while the neck is moved to restore normal function and reduce discomfort. Target muscles include the pectoralis major, upper trapezius, levator scapulae, rhomboids, deep neck flexors, and serratus anterior.

The intervention will also include a structured exercise program designed to stretch and strengthen the neck and shoulder muscles, reduce tension, and enhance posture. Stretches will consist of sitting chair stretch, Brugger's stretch, wall angles, and doorway stretches. Strengthening activities such as the Kibler squeeze and head/neck retractions will also be incorporated. The home program will begin with gentle neck stretches, such as tilting the head toward one shoulder and holding the position for 20-30 seconds, repeating three times on each side. Chin tucks will be performed by gently retracting the chin without tilting the head, holding for 5 seconds, and repeating 10 times for 2-3 sets. These exercises aim to relieve muscle tightness, improve alignment, and help alleviate headache symptoms.

ELIGIBILITY:
Inclusion Criteria:

* * Aged between 20-50 years

  * Both Male and females
  * Individuals diagnosed with neck pain accompanied by headaches.
  * Individuals with Unilateral or Bilateral cervicogenic headache.
  * Headache at least 3 times during the last 3 months.

Exclusion Criteria:

* * History of inflammatory disorders (e.g Rheumatoid Arthritis).

  * History of trauma to the cervical region.
  * History of Neurological conditions (myelopathy, radiculopathy or disc problems).
  * Taking medications for headache.
  * Pregnancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) score | Baseline, 4 weeks, and 8 weeks after start of intervention
  The purpose of the Neck Disability Index (NDI) questionnaire is to gather data on how your neck pain has impacted your capacity to function in daily life. The NDI is divided into ten categories, each of which is rated from 0 to 5, where 5 represents "worst imaginable pain" and 0 represents "no pain". The sum of the points determines the final score, with 0 denoting no activity constraints and 50, or 100%, denoting entire activity limitations.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) score. | Baseline, 4 weeks, and 8 weeks after start of intervention
  In the segmented numerical version of the NPRS, a respondent chooses a whole number (0-10 integers) that most accurately represents the level of pain they are experiencing. A horizontal bar or line is the standard format. It takes less than a minute to finish the NPRS. Greater pain intensity is indicated by higher scores, which range from 0 to 10.
Headache Disability Index (HDI) score | Baseline, 4 weeks, and 8 weeks after start of intervention
  The Henry Ford Hospital Headache Disability Inventory/Index (HDI) was created to measure how headaches affect day to day functioning. A 25-item headache questionnaire that was developed from the case history answers of individuals who had headaches was divided into functional and emotional subscales to evaluate how headaches and their management affected daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- The University Of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No